CLINICAL TRIAL: NCT00263016
Title: A Phase II Pilot Study of Combination of Irinotecan and Cisplatin in Docetaxel/Cisplatin-Responsive Advanced Non-Small Cell Lung Cancer
Brief Title: Docetaxel in Non Small Cell Lung Cancer (NSCLC)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow recruitment
Sponsor: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XRP6976B_2503
Record Dates: First submitted 2005-12-06; First posted 2005-12-07 (Estimated); Last update posted 2008-03-20 (Estimated); Status verified 2008-03

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Docetaxel

INTERVENTIONS:
Drug: Docetaxel

SUMMARY:
Primary Objective:

* To compare the tumour response rate of combination chemotherapy irinotecan/cisplatin (IC) versus docetaxel/cisplatin (DC) in advanced NSCLC patients who responded to 3 courses of docetaxel/cisplatin.

Secondary Objectives :

* To compare the time to progression after chemotherapy treatment between the IC and DC arms of treatment.
* To compare the toxicity profile of the IC and DC arms of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven non-small cell lung carcinoma at first diagnosis.
* Stage IIIB or IV disease.
* Tumour considered unresectable.
* Performance status Karnofsky index > 60% or WHO performance status < or = 1.
* Previous therapy

  * Chemotherapy: None.
  * Previous radiation therapy: prior irradiation for NSCLC is permitted, however, the measurable or evaluable non-measurable disease must be completely outside the radiation portal.
* Laboratory requirements:

  * Hematology:

    * Neutrophils ≥ 2.0 10^9/l,
    * Platelets ≥ 100 10^9/l,
    * Hemoglobin ≥ 10 g/dl.
  * Hepatic function:Total bilirubin < 1 Upper Normal Limit (UNL), AST (SGOT) and ALT (SGPT) < 2.5 UNL,Alkaline phosphatase < 5 UNL ; except in presence of only bone metastasis and in absence of any liver disorders. Patients with AST and/or ALT > 1.5 x UNL associated with alkaline phosphatase > 2.5 x UNL are not eligible for the study.
  * Renal function: Creatinine < 140 µmol/l (1.6 mg/dl) ; if limit values, the calculated creatinine clearance should be > 60 ml/min.

Exclusion Criteria:

* Pregnant, or lactating patients; patients of childbearing potential must implement adequate contraceptive measures during study participation.
* Known clinical brain or leptomeningeal involvement.
* Pre-existing motor or sensory neurotoxicity of a severity > grade 1 by National Cancer Institute criteria.
* Other serious illness or medical condition:

  * Congestive heart failure or unstable angina pectoris even if it is medically controlled. Previous history of myocardial infarction within 1 year from study entry, uncontrolled hypertension or high risk uncontrolled arrhythmias.
  * History of significant neurologic or psychiatric disorders including psychotic disorders, dementia or seizures that would prohibit the understanding and giving of informed consent.
  * Active uncontrolled infection.
  * Peptic ulcer, unstable diabetes mellitus or other contraindication for the use of corticosteroids.
* Past or current history of neoplasm other than non-small cell lung cancer, except for curatively treated non-melanoma skin cancer, in situ carcinoma of the cervix.
* Concurrent treatment with prednisone (or equivalent) except as use for the prophylactic medication regimen, treatment of acute hypersensitivity reactions, treatment of nausea / vomiting or unless chronic treatment (initiated > 6 months prior to study entry) at low dose (< 20 mg methylprednisolone or equivalent).
* Definite contraindications for the use of corticosteroids.
* Concurrent treatment with other experimental drugs. Participation in another clinical trial with any investigational drug within 30 days prior to study entry.
* Concurrent treatment with any other anti-cancer therapy.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2005-05

PRIMARY OUTCOMES:
Tumour response rate
Survival at 1 year

SECONDARY OUTCOMES:
Time to progression

CONTACTS AND LOCATIONS:
Overall Officials: Iris CHAN, MD, Study Director — Sanofi
Locations (1):
- Sanofi-aventis, Hong Kong, Hong Kong